CLINICAL TRIAL: NCT02152618
Title: Permanency Innovations Initiative- Kansas Intensive Permanency Project
Brief Title: Kansas Intensive Permanency Project
Acronym: PIIKIPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Westat (Other)
Collaborators: Children's Bureau ACYF (Unknown); Office of Planning, Research & Evaluation (U.S. Federal Agency); University of Kansas School of Social Welfare (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HHSP23320095655WC-KS
Record Dates: First submitted 2014-04-14; First posted 2014-06-02 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Serious Emotional Disturbance; In Foster Care
Keywords: Serious emotional disturbance; foster care; child protective services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Other: Parent Management Training - Oregon Model (PMTO)
- Comparison (No Intervention)

INTERVENTIONS:
Other: Parent Management Training - Oregon Model (PMTO) — Evidence-based, behavioral parent management training model, Parent Management Training - Oregon Model (PMTO) tailored to address permanency barriers of parents of children with SED.
  Arms: Treatment

SUMMARY:
The intervention provides services to children with Serious Emotional Disturbance (SED) who are in foster care and to their parent(s) to prepare the families for reunification.

DETAILED DESCRIPTION:
The intervention provide services to children with Serious Emotional Disturbance (SED) who are in foster care and to their birth parents to prepare the families for reunification. The evaluation follows a randomized design. The pretest will assess the procedures and instruments for collecting data on child, youth, and family functioning. Ultimately, after the pretest is complete, the data collected through the evaluation will provide information on the extent to which the intervention achieved its goal of improving parenting skills and enhancing readiness for reunification among the families who received the services.

ELIGIBILITY:
Inclusion Criteria:

* Children age 3-16 with severe emotional disturbances
* In foster care and their families (parents).

Exclusion Criteria:

-

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1652 (Actual)
Dates: Start 2010-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Time to stable permanence | Measured from the date of random assignment to the discharge date or to the end of the study period for cases that did not discharge
  Measured by administrative data from the Adoption and Foster Care Analysis and Reporting System (AFCARS)
Positive parenting behaviors | Pre intervention, post intervention and at 12-months
  Measured by administering two standardized instruments: 1) the Caregiver Wish List (CWL); and, 2) the Family Interaction Task (FIT).

SECONDARY OUTCOMES:
Use of community resources & social supports | Pre intervention, post intervention and at 12-months
  Measured by observing the results of a subscale of a standardized instrument, the North Carolina Family Assessment Scale, General and Reunification services (NCFAS-G+R). The subscale is identified as "social/community life."
Readiness for Reunification | Pre intervention, post intervention and at 12-months
  Measured by the "readiness for reunification" subscale of the North Carolina Family Assessment Scale, General and Reunification services (NCFAS-G+R).
Improve parent mental health & Substance Abuse | Pre intervention, post intervention and at 12-months
  Measured by the relevant items on the North Carolina Family Assessment Scale, General and Reunification services (NCFAS-G+R).
Child behavior | Intake & every 6-months post intake
  Measured with Social Skills Improvement System rating scales (SSIS).
Child functioning | Intake & every 6-months post intake
  Measured by assessing the child's functioning with the Child and Adolescent Functional Assessment Scale (CAFAS) for school-aged children and the Preschool and Early Childhood Functional Assessment Scale (PECFAS) for preschool-aged children.
Reunification | 18 months post intervention start date
  Measured using data from Kansas' state administrative database for child welfare as reported to AFCARS/NCANDS.
Long-term foster care | Measured at 6 and 12 months post entry into foster care
  Measured by using data from Kansas' state administrative database for child welfare as reported to AFCARS/NCANDS.
Stable permanency | Measured at 6 and 12 months post entry into foster care
  Measured by using data from Kansas' state administrative database for child welfare as reported to AFCARS/NCANDS.
Child safety | Measured at 6 and 12 months post entry into foster care
  Measured by using data from Kansas' state administrative database for child welfare as reported to AFCARS/NCANDS.
Coercive parenting practices | Pre intervention, post intervention and at 12-months
  Measured by administering two standardized instruments: 1) the Caregiver Wish List (CWL); and, 2) the Family Interaction Task (FIT).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Testa, PhD., Principal Investigator — University of North Carolina; Andrea Sedlak, PhD., Study Director — Westat